CLINICAL TRIAL: NCT02250157
Title: A Dose-regimen Finding Study to Evaluate Safety, Tolerability, Pharmacokinetics and Activity of Oratecan in Subjects With Advanced Malignancies
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Athenex, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ORTE-01-14-US
Record Dates: First submitted 2014-09-22; First posted 2014-09-26 (Estimated); Last update posted 2022-02-22 (Actual); Status verified 2022-02

CONDITIONS: Solid Tumor
MeSH Terms: interventions — Irinotecan; 4-oxo-4H-chromene-2-carboxylic acid (2-(2-(4-(2-(6,7-dimethoxy-3,4-dihydro-1H-isoquinolin-2-yl)-ethyl)-phenyl)-2H-tetrazol-5-yl)-4,5-dimethoxyphenyl)amide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Part 1 (Experimental): Part 1 of this study is a "3+3" design to define the MTD of Oratecan in up to 60 evaluable subjects. It will be conducted in 2 parts; 1A will test the oral liquid formulation and 1B will test the oral tablet formulation of irinotecan.
  Interventions: Drug: Oratecan
- Part 2 (Experimental): Part 2 will enroll an additional 10 subjects at the Part 1 MTD to further characterize the safety, tolerability, pharmacokinetics, and activity of Oratecan at that dose.
  Interventions: Drug: Oratecan

INTERVENTIONS:
Drug: Oratecan
  Other Names: Camptosar, HM30181

SUMMARY:
This study a nonrandomized, open-label, uncontrolled, single group assignment, safety and activity study in subjects with histologically or cytologically confirmed solid tumor that is metastatic or unresectable and for which standard curative or palliative measures do not exist or are no longer effective.

DETAILED DESCRIPTION:
This study consists of Part 1 and Part 2. Part 1 of this study is a "3+3" design to define the MTD of Oratecan in up to 60 evaluable subjects. It will be conducted in 2 parts; 1A will test the oral liquid formulation and 1B will test the oral tablet formulation of irinotecan. Part 2 will enroll an additional 10 subjects at the Part 1 MTD to further characterize the safety, tolerability, pharmacokinetics, and activity of Oratecan at that dose.

Irinotecan (CPT-11) is a potent anticancer drug under the class of camptothecins that is marketed under the trade name Camptosar. Irinotecan is a prodrug that is activated via carboxylesterase in liver and intestines to its active form, SN38 which is approximately 1000 times more cytotoxic than irinotecan itself.

The investigational product (IP) Oratecan is comprised of the approved drug irinotecan with HM30181 methanesulfonate monohydrate (HM30181), a novel p-glycoprotein (P-gp) pump inhibitor. Oratecan is intended for the treatment of irinotecan-responsive cancers. The antitumor activity of Oratecan is due to the action of irinotecan. Combining HM30181 with irinotecan allows intestinal absorption and systemic exposure of irinotecan and its active metabolite, SN38, at therapeutic levels after oral administration.

ELIGIBILITY:
Inclusion Criteria:

* Signed written informed consent.
* ≥ 18 years of age.
* Histologically or cytologically confirmed solid tumor that is metastatic or unresectable and for which standard curative or palliative measures do not exist or are no longer effective.
* Measurable disease as per Response Evaluation Criteria in Solid Tumors (RECIST) Version 1.1 criteria.
* Adequate bone marrow reserve as demonstrated by :
* Absolute Neutrophil Count (ANC) ≥ 1.5 x 10⁹/L.
* Platelet count ≥ 100 x 10⁹/L.
* Hemoglobin ≥ 9 g/L.
* Adequate liver function as demonstrated by:
* Total bilirubin of ≤ 1.5 mg/dL or ≤ 2.0 mg/dL for subjects with liver metastasis.
* Alanine aminotransferase ≤ 3 x ULN or ≤ 5 x ULN if liver metastasis is present.
* Alkaline phosphatase ≤ 3 x ULN or ≤ 5 x ULN if bone metastasis is present
* Adequate renal function as demonstrated by serum creatinine ≤ 1.5 x ULN or 24-hour urine creatinine clearance calculation ≥ 60 mL/min.
* Eastern Cooperative Oncology Group performance status of 0 to 1.
* Life expectancy of at least 3 months.
* Woman must be postmenopausal (> 12 months without menses) or surgically sterile (ie, by hysterectomy and/or bilateral oophorectomy) or must be using effective contraception (ie, oral contraceptives, intrauterine device, double barrier method of condom and spermicide) and agree to continue use of contraception for 30 days after their last dose of IP.
* Sexually active male subjects must use a barrier method of contraception during the study and agree to continue the use of male contraception for at least 30 days after the last dose of IP.

Exclusion Criteria:

* Subjects who are homozygous for the UGT1A1*28 allele
* Have not recovered to ≤ Grade 1 toxicity from previous anticancer treatments or previous IPs.
* Received IPs within 14 days or 5 half-lives of the first study dosing day, whichever is longer.
* Are currently receiving other medications intended for the treatment of their malignancy.
* Women who are pregnant or breast feeding.
* Taking a medication known to be clinically significant P-gp inhibitors or inducers within 14 days of treatment with Oratecan.
* Chronically taking an oral medication known to be a P-gp substrate within 7 days of starting treatment with Oratecan.
* Taking a medication known to be a clinically significant cytochrome (CYP) 3A4 strong inhibitor (eg, ketoconazole within 14 days) or strong inducers (eg, rifampin and St. John's Wort within 14 days) of starting treatment with Oratecan. http://www.fda.gov/Drugs/DevelopmentApprovalProcess/DevelopmentResources/DrugInteractionsLabeling/ucm080499.htm
* Require therapeutic use of anticoagulation medications
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, myocardial infarction within the last 6 months, unstable angina pectoris, cardiac arrhythmia, chronic pulmonary disease requiring oxygen, known bleeding disorders, or any concomitant illness or social situation that would limit compliance with study requirements.
* Major surgery to the upper gastrointestinal (GI) tract, or have a history of GI disease or other medical condition that, in the opinion of the investigator may interfere with oral drug absorption.
* Allergy or sensitivity to irinotecan or cranberry-grape juice, or any of the irinotecan tablet excipients. .

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2014-09-05 (Actual); Primary Completion 2020-03-04 (Actual); Study Completion 2020-03-04 (Actual)

PRIMARY OUTCOMES:
Number of participants with dose limiting toxicities | 2 years

SECONDARY OUTCOMES:
Number of patients with adverse events | 2 years
Area under the plasma concentration versus time curve | 2 years
  Determine the amount of Oratecan in participants blood (pharmacokinetics)
Tumor measurements per RECIST 1:1 | 2 years
  Assess preliminary anti-tumor activity

CONTACTS AND LOCATIONS:
Overall Officials: Donal Landers, MD, Study Chair — Athenex, Inc.
Locations (2):
- United States (2):
  - University of Colorado Cancer Center, Aurora, Colorado
  - Roswell Park Cancer Institute, Buffalo, New York